CLINICAL TRIAL: NCT03239002
Title: Antenatal Detection by Array CGH Genomic Rearrangements Unbalanced Front Uninsulated Thick Neck or a Combination of Two Signs of Ultrasound Calling Normal Karyotype
Acronym: CGH Array
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2010_24; 2011-A00105-36 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-07-31; First posted 2017-08-03 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Abnormality of the Neck; Fetus; Abnormal, Affecting Management of Pregnancy
MeSH Terms: conditions — Antisocial Personality Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is the first study with a real diagnostic and prognostic focus in prenatal. In addition to this innovative aspect, the identification of cryptic imbalances in fetuses with malformative syndrome would be an invaluable resource for the identification of new genes involved in development, as is already the case for postnatal studies.

This research aims to:

1. to test the feasibility of this protocol, ie the practical application of this new technology in the context of prenatal diagnosis,
2. demonstrate and evaluate the possible involvement of cryptic chromosomal abnormalities in fetuses with a thick neck associated with other malformations and recruited on the strict criteria mentioned above,
3. assist in the diagnosis of these fetuses and genetic information for their families,
4. identify new regions of the genome potentially involved in the occurrence of congenital malformations.

ELIGIBILITY:
Inclusion Criteria:

* a karyotype performed from a trophoblast biopsy or an amniotic fluid puncture is normal or apparently balanced.
* The fetuses included in the study should have one of the following two criteria:
* 1) Thick bone (greater than 99th percentile, between week 11 and week 13 of amenorrhoea plus 6 days, correlated to a cranio-caudal length measured between 45 and 84 mm) detected in the first trimester of pregnancy associated with One or more echographic sign (s).
* 2) At least two ultrasound call signs involving the following organs (heart, kidney, brain, limbs, digestive tract, face) or intrauterine growth retardation (less than 3rd percentile) associated with one of these Signs of appeal.

Exclusion Criteria:

* The parturientes in emergency situation,
* Benefiting from a legal protection (guardianship / curatorship)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 200 parturientes aged 18 to 45 years
Study Population: the parturients aged 18 to 45 years for whom a karyotype performed from a trophoblast biopsy or amniotic fluid puncture is normal or apparently balanced
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-07; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of patient with Ultrasound call signs (thick neck and / or any other organ concerned) | During the first trimester of pregnancy

SECONDARY OUTCOMES:
CGH-array analysis | During the first trimester of pregnancy
  CGH-array result: normal, deletion or duplication, de novo or inherited, size, type and number of genes involved

CONTACTS AND LOCATIONS:
Overall Officials: Véronique HOUFFLIN-DEBARGE, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Jeanne de Flandre - CHRU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No